CLINICAL TRIAL: NCT02264756
Title: Evaluating the Effectiveness of an Antimicrobial Stewardship Program on Reducing the Length of Stay of Immune-competent Adult Patients Admitted to a Hospital Ward With a Diagnosis of Community-acquired Pneumonia
Brief Title: Improving Antibiotic Use in Hospitalized Patients With Pneumonia
Acronym: CAPASP
Status: Completed | Type: Observational
Sponsor: Giulio DiDiodato (Other)
Responsible Party: Sponsor-Investigator, Giulio DiDiodato, Medical Lead, Antimicrobial Stewardship Program, Royal Victoria Hospital, Canada
Organization: Royal Victoria Hospital, Canada (Other)
Other Study IDs: CAPASP2013
Record Dates: First submitted 2014-09-30; First posted 2014-10-15 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Pneumonia
Keywords: Community-acquired pneumonia; Pragmatic clinical trial; Antimicrobial stewardship; length of stay; stepped-wedge design; time-dependent bias
MeSH Terms: conditions — Pneumonia; Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ward CAP: Adult immune-competent patients admitted to ward with clinical diagnosis of community-acquired pneumonia will be potentially exposed to ASP review
  Interventions: Other: ASP review

INTERVENTIONS:
Other: ASP review — patients admitted to hospital with a diagnosis of community-acquired pneumonia will be reviewed by team members of antimicrobial stewardship program and subsequently feedback to attending physicians will be offered in the form of recommendations for antibiotic management
  Other Names: prospective chart audit and attending physician feedback

SUMMARY:
The purpose of the study is to determine whether an antimicrobial stewardship program can decrease the length of hospital stay for patients with pneumonia. The antimicrobial stewardship program is run by a pharmacist and doctor with extensive training in managing infectious diseases. These two health care professionals are responsible for reviewing the records of patients admitted to hospital with pneumonia, and then making specific recommendations to the patient's attending physician about how to manage antibiotic treatment. These recommendations might include discontinuing the antibiotic, or changing the way antibiotics are delivered from intravenous form to pill form, among many other potential options. The attending physician considers whether these recommendations should be followed or rejected. The study has a control group of patients who are not reviewed by the antimicrobial stewardship team, and their length of hospital stay will be compared to the reviewed group of patients. Any differences between these two groups will be assumed to be due to the impact of the antimicrobial stewardship program. So far, no previous study has been able to demonstrate that an antimicrobial stewardship program can reduce the length of stay of patients admitted to hospital with pneumonia. This study has some important differences from previous studies that may make its conclusions more accurately reflect the true impact of antimicrobial stewardship programs. The most important difference is how the timing of the review is modelled in the analysis of the study results. Because the timing of the review varies between patients, with some patients being reviewed at earlier and some at later times, this subtle difference, if not accounted for in the analysis, can mask a true positive effect of the program on length of stay. The investigators study will account for this variation.

DETAILED DESCRIPTION:
In immune-competent adult patients admitted to a hospital ward with a diagnosis of community-acquired pneumonia, does a multi-faceted ASP utilizing prospective chart audit and feedback compared with usual care reduce the LOS without increasing the risk of death or readmission at 30 days post-discharge from hospital? In Ontario, pneumonia is the leading cause of death from bacterial infections and accounts for over 18,000 years of life lost annually due to premature mortality. Pneumonia accounts for the majority of antibiotic utilization in both hospital and outpatient settings. Evidence-based guidelines for the diagnosis and management of pneumonia are available to physicians. Adherence to these evidence-based guidelines is associated with both reduced mortality and antibiotic utilization.

Antimicrobial stewardship is defined as any intervention that minimizes unwarranted variation in antimicrobial utilization from evidence-based best practice with the intent of improving patient safety and quality of care. Unwarranted refers to the absence of patient- or disease-specific reasons to justify practice variation from evidence-based practice standards. Antimicrobial stewardship can be operationalized in many different ways, but prospective audit and feedback (persuasive approach) and restricted antimicrobial prescribing policies (restrictive approach) appear to be the most efficacious interventions to achieve the goals of antimicrobial stewardship. Antimicrobial stewardship programs have demonstrated efficacy in improving antimicrobial prescribing and reducing rates of hospital-acquired infections. Antimicrobial stewardship programs directed to CAP patients have demonstrated reductions in mortality, but have failed to demonstrate reductions in length of stay.

All participants will be admitted patients to the Royal Victoria Regional Health Centre (RVRHC), a 319 bed community-based, university-affiliated, acute care hospital located in Barrie, Ontario, Canada.

All patients enrolled in the study will be admitted to one of four medical wards. All study patients will be admitted to a hospitalist service. Admission to any medical ward is controlled by bed allocation, a non-medical administrative service within the hospital responsible for patient flow and assigning patient care. Hospitalists are not assigned to any one specific medical ward, but provide care across all medical wards.

All eligible CAP who meet the ASP review criteria will be exposed to the ASP intervention. The ASP intervention (ASP-i) consists of a prospective chart audit and physician feedback (persuasive) approach . The ASP members who conduct all the audits and make recommendations consist of an infectious diseases-trained pharmacist (LM) and an infectious diseases trained physician (GD). All patients are reviewed by both members. The ASP intervention (ASP-i) recommendations are guided by the Infectious Diseases Society of America CAP guidelines and the Canadian Thoracic Society guidelines for the management of chronic obstructive pulmonary disease. The possible ASP-i recommendations are based on those recommended by the National Health Service in the United Kingdom and include the following:

i) No change to current care ii) Discontinue antibiotic(s) iii) Intravenous to oral conversion iv) Duration of therapy v) Dosing change vi) Narrow or broaden spectrum of therapy The ASP-i recommendations are not mutually exclusive. All recommendations are documented in the patient's electronic medical record and communicated directly to the attending physician by the ASP members.

This is a pragmatic controlled clinical study intended to measure the effectiveness of a 'real world' program. The ASP-i will be implemented in a modified stepped wedge design; baseline patient data will be collected for all enrolled patients on each of the medical wards for the first three months of the study, and then the ASP-i will be introduced to each medical ward in a non-randomized sequential fashion in two month intervals until all medical wards are exposed to the intervention.

The unit of analysis will be individual patients adjusted for potential clustering effects within hospital wards.

The primary outcome is length of hospital stay (LOS) measured in minutes from the documented time of admission to the documented time of discharge (or censoring). All patients will be administratively censored at 14 days after hospital admission if they have not been discharged home.

Enrollment of patients started on April 1, 2013. The study is expected to enroll patients until March 31, 2015. All consecutive patients that meet the inclusion criteria and have no exclusion criteria will be eligible for the intervention. The ASP-i intervention may be implemented anytime after 48 hours post-admission in those patients who meet the criteria for ASP review. All patients who have not experienced an outcome at 14 days after admission will be censored from the study. Patients who die or are transferred from the ward (to the intensive care unit or other hospital) will also be censored. Patients who are discharged from hospital and are not censored will be contacted at 30 days post-discharge to determine their adherence with antibiotic prescription (if relevant), survival status and readmission status.

The sample size expected for the current study is 'fixed' and has been previously estimated to be between 400 to 500 CAP patients per calendar year. The accrual period will be 24 months. Assuming 70% of patients in the control arm will achieve the primary outcome of being discharged alive from hospital, and setting power = 0.8 and statistical significance (2-sided) α = 0.05, the detectable ASP-i effect size is estimated to be up to an approximately 20% reduction in length of stay.

An extended Cox regression analysis will be used to compare the primary and secondary outcomes between the control and intervention groups. Violations of the proportional hazards assumption for each covariate will be identified by using the method of Schoenfeld residuals. Results will be reported as hazard ratios with 95% confidence intervals. Time to ASP-i will be modeled as a time-variant covariate in the final model to account for any time-dependent bias.

Other variables known to be associated with the primary and secondary outcomes will also be included in the final model, and include; age, sex, charlson comorbidity index, CURB-65 score, time (days) to clinical resolution, and complications from pneumonia such as empyema. Fixed effects of wards on the outcomes will accounted for by including them as indicator variables in the final model. Maturation of ASP-i effect on outcomes over time will be adjusted by including a categorical time variable in the final model (time variable will be defined as 'quarter' from start of study). A dichotomous variable for acceptance or rejection of the ASP-i will be part of an interaction term with the control/intervention group variable to permit a per protocol analysis.

ELIGIBILITY:
Inclusion Criteria:

* have a positive Febrile Respiratory Illness (FRI) screen on admission to hospital (http://www.health.gov.on.ca/fr/public/programs/emu/sars/reports/dir_122303_acute_care_nonoutbreak.pdf)
* diagnosed with pneumonia by the admitting physician (Acute exacerbations of chronic obstructive lung disease are considered within the definition of pneumonia for the purposes of this study as they are commonly treated with the same antimicrobial regimens as patients with pneumonia)
* admitted to a medical ward

Exclusion Criteria:

* hospitalized for ≥ 48 consecutive hours in the preceding 3 months
* receiving immunosuppressants [defined as ≥ 40 mg prednisone daily (or steroid equivalent) for ≥ 2 weeks preceding hospitalization OR any other immunosuppressant used for systemic illness OR to prevent transplant rejection]
* neutropenic [defined as a polymorphonuclear count ≤ 0.5 x 109 cells/L] from any cause
* immunocompromised [defined as having leukemia, lymphoma, HIV with CD4 cell count ≤ 200, splenectomy or on cytotoxic chemotherapy]
* admitted to high acuity units such as intensive care units
* require mechanical ventilation, either non-invasive or invasive
* have a life expectancy of ≤ 3 months (palliative)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult immune-competent hospital inpatients admitted to a ward at the Royal Victoria Regional Health Centre, Barrie, Ontario, Canada
Sampling Method: Non-Probability Sample
Enrollment: 763 (Actual)
Dates: Start 2013-04; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Hospital length of stay | Patients will be followed for 14 days from date of admission and if not discharged will be administratively censored
  Time to discharge or censoring event

SECONDARY OUTCOMES:
30-day post-discharge mortality rate | 30 calendar days after hospital discharge
  all cause mortality at 30 days post-discharge from hospital
30-day post-discharge readmission rate | 30 calendar days after hospital discharge
  all cause readmission rate at 30 days post-discharge from hospital
Days of antimicrobial therapy | Total days of antimicrobial therapy for each antibiotic calculated from date of first administration on admission to hospital to date of discontinuation (or to date of censoring, whichever comes first) upto a maximum of 30 days post-discharge follow-up
  Total days of antimicrobial therapy used per patient upto a maximum of 30-days post-discharge from hospital
Duration of antimicrobial therapy | Total duration of all antibiotics administered starting from date of administration of first antibiotic to date of discontinuation of last antibiotic (or to date of censoring, whichever comes first) upto a maximum of 30 days post-discharge from hospital
  Total duration of antimicrobial therapy per patient upto a maximum of 30-days post discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Giulio DiDiodato, MD, Principal Investigator — Royal Victoria Regional Health Centre
Locations (1):
- Royal Victoria Regional Health Centre, Barrie, Ontario, Canada

REFERENCES:
- [Derived] DiDiodato G, McArthur L, Beyene J, Smieja M, Thabane L. Can an antimicrobial stewardship program reduce length of stay of immune-competent adult patients admitted to hospital with diagnosis of community-acquired pneumonia? Study protocol for pragmatic controlled non-randomized clinical study. Trials. 2015 Aug 14;16:355. doi: 10.1186/s13063-015-0871-2. PMID 26272324